CLINICAL TRIAL: NCT05204927
Title: A Multi-Center, Open-Label, Randomized Phase 3 Trial Comparing the Safety and Efficacy of 177Lu-PSMA-I&T Versus Hormone Therapy in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: 177Lu-PSMA-I&T for Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Curium US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CURLu177PSM0001
Record Dates: First submitted 2021-12-01; First posted 2022-01-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Metastasis From Malignant Tumor of Prostate
Keywords: Radioligand Therapy; Prostate Cancer; 177Lu-PSMA; PSMA; ECLIPSE
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Prednisone; enzalutamide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized on a 2:1 basis to receive Lu177-PSMA (Investigational Arm) or standard of care hormone therapy (Control Arm). The Control Arm will consist of treatment with either abiraterone with prednisone or enzalutamide depending on the clinical judgement of the investigator. Participants who are randomized to the control arm who demonstrate radiographic progression may be eligible to crossover to receive Lu177-PSMA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Of Care Hormone Therapy (Active Comparator): Abiraterone with Prednisone or Enzalutamide
  Interventions: Drug: Abiraterone with Prednisone or Enzalutamide
- Investigational Drug (Experimental): 177Lu-PSMA-I&T
  Interventions: Drug: 177Lu-PSMA-I&T

INTERVENTIONS:
Drug: 177Lu-PSMA-I&T — Radioligand therapy
  Arms: Investigational Drug
Drug: Abiraterone with Prednisone or Enzalutamide — Hormone Therapy
  Arms: Standard Of Care Hormone Therapy

SUMMARY:
A Multi-Center, Open-Label, Randomized Phase 3 Trial Comparing the Safety and Efficacy of 177Lu-PSMA-I&T versus Hormone Therapy in Patients with Metastatic Castration-Resistant Prostate Cancer.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, randomized, Phase 3 study evaluating Lutetium 177Lu-PSMA-I&T as treatment compared to standard of care hormone therapy in men with metastatic Castration-Resistant Prostate Cancer.

The study will include a total of 400 patients with metastatic prostate cancer and documented positive PSMA PET imaging. Patients will be randomized at a ratio of 2:1 to receive either 177Lu-PSMA-I&T or hormone therapy (abiraterone or enzalutamide) respectively. Patients randomized to the investigational product will receive up to 6 treatments every 6 weeks at a dose of 200 mCi (7.4 GBq). All patients will be followed for adverse events and safety labs throughout the course of the study. Progression of disease will be assessed radiographically using Prostate Working Group Criteria 3 (PWGC3) and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of conventional imaging as well as PSA levels and symptom recording throughout the course of treatment.

30 patients will participate in a pharmacokinetic and radiation dosimetry sub-study at selected participating clinical sites. Sub-study participants will receive SPECT imaging after each treatment cycle for dosimetry analysis. Sub-study participants will not be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18 years or older able to understand and provide signed written informed consent.
2. Histologically or pathologically confirmed prostate adenocarcinoma without predominant small cell component.
3. Progressive disease by one or more of the following criteria:

   1. Serum/plasma PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week apart with a minimum start value of >2 ng/mL.
   2. Progression of measurable disease (RECIST 1.1) or presence of at least two new bone lesions (PCWG3 criteria).
4. Previous treatment with next-generation androgen receptor (AR)-directed therapy (e.g. abiraterone, enzalutamide, apalutamide, darolutamide).

   1. Must have received no more than one previous AR-directed therapy.
   2. Must have been administered ARAT (abiraterone, enzalutamide, darolutamide, or apalutamide) in the castration-sensitive or castration-resistant setting.
   3. Must have progressed while on ARAT.
5. PSMA-PET scan (e.g., 68Ga-PSMA-11 or 18F-DCFPyL) positive as determined by central reader.
6. Effective castration with serum testosterone level of <50 ng/dL and plan to continue with chronic medical or surgical castration.
7. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
8. Patients with HIV that are healthy and with a low risk of acquired immune deficiency syndrome related outcomes may participate in the trial at the investigators' discretion.
9. Patients with HBV and HCV may also participate if symptoms are sufficiently managed.
10. Life expectancy of at least 6 months as assessed by investigator.
11. Willing to initiate ARAT therapy determined by investigator.
12. For patients who have partners of childbearing potential: The patient and/or partner must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 6 months after the last study drug administration.

Exclusion Criteria:

1. Prior treatment with radioligand therapy including other lutetium-labeled compounds.
2. Prior treatment with radium-223 (Xofigo) within the past 12 weeks.
3. Prior chemotherapy treatment for castration-resistant prostate cancer. Prior docetaxel use in the hormone-sensitive setting is permitted, as long as no more than 6 doses were received, the last dose was administered >1 year prior to consent, and disease progression did not occur during docetaxel treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≥ 2
5. Patients with known HRR gene-mutation (BRCA 1/2 encompassing both germline and somatic) who have not been previously treated with olaparib or rucaparib.
6. Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
7. Inadequate organ and bone marrow function as evidenced by:

   1. Hemoglobin < 8 g/dL.
   2. Absolute neutrophil count < 1.5 x 109/L.
   3. Platelet count < 100 x 109/L.
   4. AST/SGOT and/or ALT/SGPT > 3.0 x ULN.
   5. Total bilirubin > 2 x ULN unless patient has known Gilbert's syndrome and then may be 3 x ULN.
   6. Creatinine clearance (CrCl) < 50 mL/min based on the Cockcroft-Gault equation.
   7. Albumin ≤ 2.75 g/dL
8. Patients who undergo a transfusion for the sole purpose of meeting eligibility for this trial will be excluded.
9. Assessment by the Investigator as unable or unwilling to comply with the requirements of the protocol.
10. Use of an investigational therapeutic drug within the last 4 weeks prior to start of study treatment or scheduled to receive one during the study period.
11. Known CNS metastasis unless received therapy, asymptomatic and neurologically stable.
12. Patients receiving zoledronic acid for bone-targeted therapy must be on stable dose for 4 weeks prior to randomization.
13. Major surgery within 30 days of randomization as determined by the Investigator.
14. Patients with active significant cardiac disease defined by any of the following:

    1. New York Heart Association class 3 or 4 congestive heart failure within 6 months of signing the ICF unless treated with improvement.
    2. Current diagnosis of electrocardiogram abnormalities with significant cardiac arrhythmias
    3. History of long QT syndrome or know history of Torsades de Pointe
    4. History of myocardial infarction, angina pectoris, or coronary artery bypass graft within 6 months of ICF signature
15. Participants with symptomatic cord compression or clinical/radiological findings indicating impending spinal cord compression
16. Patients with a superscan seen on baseline bone scan as determined by investigator.
17. Active malignancy other than low-grade non-muscle-invasive bladder cancer and non-melanoma skin cancer
18. Previous use of G-CSF for persistent neutropenia after standard of care treatment.
19. Participants who have a pregnant partner or are capable of fathering a child and who are unwilling to take precautions to prevent potential harm to the fetus or prevent pregnancy.
20. Participants with active Covid19. Recovered patients may be included when completely recovered (no symptoms at least 28 days before study medication and a negative Covid test within 72 hours).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 439 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival | 34 weeks
  Radiographic progression free survival (rPFS), defined as the time from randomization to radiographic progression (using PCWG3 and RECIST 1.1 criteria as assessed by blinded independent central review [BICR]) or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 156 weeks
  Time (weeks) from randomization to death due to any cause.
Second Radiographic Progression Free Survival (rPFS 2) | 156 weeks
  Time from randomization to the second radiographic progression or death in participants who crossover.
Progression Free Survival | 156 weeks
  First occurrence of PCWG3 progression, clinical/symptomatic progression and/or pain progression, or death due to any cause.
Second Progression-Free Survival | 156 weeks
  Second occurrence of PCWG3 progression, clinical/symptomatic progression and/or pain progression, or death due to any cause.
PSA50 Response Rate | 156 weeks
  Response rate of patients who achieve a reduction of ≥50% in PSA from the baseline PSA assessment.
Time to First Symptomatic Skeletal Event (SSE) | 156 weeks
  Occurrence of either bone-directed radiotherapy to relieve bone pain, new symptomatic pathologic fractures, spinal cord compression, or tumor-related orthopedic surgery.
Time to Soft Tissue Progression (STP) | 156 weeks
  Occurrence of radiographic progression in soft tissue.
Time to Chemotherapy (TTC) | 156 weeks
  Time from randomization to the initiation of chemotherapy or death.
Quality of Life Questionnaire- EORTC QLQ-C30 | 22 weeks
  The Quality of Life (QoL) will be assessed via European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30). The EORTC QLQ-C30 is a questionnaire of thirty quality of life (QoL) questions developed to assess the QoL of cancer patients. The EORTC QLQ-C30 comprises 30 items, 24 of which are aggregated into nine multi-item scales, which are scored from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (52):
- United States (37):
  - Arizona Institute of Urology, PPLC, Tucson, Arizona
  - Providence Medical Foundation, Fullerton, California
  - Long Beach Memorial Center, Long Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - San Francisco VA Health Care System, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Providence Saint John's Health Center, Santa Monica, California
  - GenesisCare USA, Boca Raton, Florida
  - Biogenix Molecular LLC, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - GenesisCare USA, Plantation, Florida
  - Florida Urology Partners, LLP, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - Kaiser Permanente Gaithersburg Medical Center, Gaithersburg, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - BAMF Health I PC, Grand Rapids, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - GenesisCare USA, Troy, Michigan
  - M Health Fairview Ridges Cancer Clinic, Burnsville, Minnesota
  - SSM Saint Louis University Hospital, St Louis, Missouri
  - Center for Clinical Theranostics Research, Washington University, St Louis, Missouri
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Central Ohio Urology Group, Gahanna, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - OHSU - Center for health and healing, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- France (8):
  - CHU Brest, Brest
  - Jean Perrin Comprehensive Cancer Center, Clermont-Ferrand
  - Institute Paoli-Calmettes, Marseille
  - Hôpital de Brabois -CHU, Nancy
  - Institut de Cancérologie de l'Ouest (ICO) St Herblain, Nantes
  - CHU Nimes, Nîmes
  - ICANS, Strasbourg
  - InstitutClaudius Regaud-IUCT-O, Toulouse
- Italy (3):
  - University Clinic Bologna, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Europeo di Oncologia (IEO) -IRCCS, Milan
- Spain (4):
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - University Hospital of Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No